CLINICAL TRIAL: NCT01607359
Title: Dabigatran Versus Warfarin Anticoagulation Before and After Catheter Ablation for the Treatment of Atrial Fibrillation
Status: Withdrawn | Type: Observational
Why Stopped: Withdrawn: It was decided not to proceed with the study at this time.
Sponsor: Corewell Health East (Other)
Collaborators: University of Pennsylvania (Other); Johns Hopkins University (Other); London Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 2007088
Record Dates: First submitted 2012-05-24; First posted 2012-05-30 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2016-12

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; dabigatran; warfarin; oral anticoagulation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- dabigatran group: All patients receiving dabigatran as periprocedural anticoagulation during the study time period
- warfarin group: A randomly selected group of patients treated with warfarin during the study time period matching the number of dabigatran treated patients in the same time period.

SUMMARY:
Both warfarin and dabigatran have been used for stroke prophylaxis at the time of catheter ablation of atrial fibrillation. Although the risks of thromboembolism and bleeding with warfarin are well established, the relative risk and benefit of dabigatran in this setting are unknown. The purposes of the study are to assess the efficacy of warfarin versus dabigatran in the prevention of stroke and other systemic embolic complications before and after catheter ablation for AF, and to compare the prevalence of serious bleeding complications with the two OAC agents.

DETAILED DESCRIPTION:
* Data from patients collected from 4 US and 1 Canadian medical center
* Retrospective record review of all patients that had undergone catheter ablation of atrial fibrillation during the time period beginning with the initiation of dabigatran therapy for stroke prophylaxis at each center and ending in November 2011.
* Dabigatran study group comprised of all patients that received dabigatran for stroke prophylaxis during the study time period.
* Warfarin comparison group to be selected from all patients that received warfarin for stroke prophylaxis during the identical study time period.
* Warfarin patients will be numbered sequentially
* A subgroup of warfarin patients identical in number to the dabigatran patients at each center will be selected using random number generator.

Patient data sets will be de-identified and compiled

* Master data set to be stored in Excel file
* Statistics to be performed with SAS (Cary, NC)
* Continuous data to be expressed as means ± S.D., compared with unpaired t-tests
* Categorical data will be compared with Fisher's exact test or Chi-square
* Complications including any thromboembolic events or any bleeding events will be recorded and the prevalence compared.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing catheter ablation for atrial fibrillation

Exclusion Criteria:

* none (retrospective trial)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing catheter ablation for atrial fibrillation
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Clinical stroke, TIA or systemic embolic complication | 30 days before or after catheter ablation
  Thromboembolic complication recorded in clinical records.
Bleeding complication | 30 days before or after catheter ablation
  Any bleeding causing additional intervention, hospitalization or pain and suffering including pericardial tamponade, large hematoma or other bleeding.

SECONDARY OUTCOMES:
Any significant complication | 30 days before or after catheter ablation
  Any significant complication that is related to the catheter ablation procedure or to the anticoagulation regimen

CONTACTS AND LOCATIONS:
Locations (1):
- Beaumont Health System, Royal Oak, Michigan, United States